CLINICAL TRIAL: NCT07285785
Title: A Randomized, Open-Label Study to Assess Pharmacokinetics of Xifaxan® 200 mg in Pediatric Subjects 6 to 11 Years of Age With Acute Diarrhea of Suspected Bacterial Etiology, and the Safety and Efficacy of Xifaxan® 200 mg Plus Oral Rehydration Therapy (ORT) Compared to ORT Alone
Brief Title: Rifaximin 200 mg Plus Oral Rehydration vs Oral Rehydration Alone in Children With Acute Diarrhea
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RFPK1991
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Diarrhea; Gastroenteritis; Bacterial Infection
Keywords: pediatric; children; rifaximin; xifaxan; Oral Rehydration Therapy (ORT); acute diarrhea; bacterial diarrhea; gastroenteritis; open-label; randomized; ages 6-11
MeSH Terms: conditions — Diarrhea; Gastroenteritis; Bacterial Infections | interventions — Rifaximin; Tablets; Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rifaximin 200 mg + ORT (Experimental): rifaximin 200 mg tablets orally three times daily for 3 days plus oral rehydration therapy (ORT) administered per investigator standard of care
  Interventions: Drug: Rifaximin 200 mg Tablet; Other: Oral Rehydration Therapy (ORT)
- ORT Alone (Active Comparator): ORT administered per investigator standard of care without rifaximin.
  Interventions: Other: Oral Rehydration Therapy (ORT)

INTERVENTIONS:
Drug: Rifaximin 200 mg Tablet — Participants receive rifaximin 200 mg tablets orally three times daily (TID) for 3 days in combination with oral rehydration therapy (ORT). Blood samples for pharmacokinetic analysis are collected on Day 1 and Day 3 at pre-dose, 1 hour post-dose, and 8 hours post-dose.
  Arms: Rifaximin 200 mg + ORT
Other: Oral Rehydration Therapy (ORT) — Participants receive oral rehydration solution according to the investigator's standard of care. This is administered either alone (for the ORT-alone arm) or in combination with rifaximin (for the rifaximin + ORT arm). Participants or caregivers complete a daily diary documenting stool frequency, stool consistency, and related symptoms.

SUMMARY:
The goal of this clinical trial is to learn how rifaximin 200 mg is processed in the body (pharmacokinetics) in children 6 to 11 years old with acute diarrhea that may be caused by bacteria. It will also learn about the safety and effectiveness of rifaximin when given with oral rehydration therapy (ORT) compared with ORT alone. The main questions it aims to answer are:

How does rifaximin 200 mg move through and leave the body in children with acute diarrhea?

Is rifaximin safe for children in this age group?

Does rifaximin plus ORT help resolve diarrhea faster than ORT alone?

Researchers will compare rifaximin plus ORT to ORT alone to see if adding rifaximin improves outcomes.

Participants will:

Take one rifaximin 200 mg tablet + ORT three times a day for 3 days or receive ORT alone

Receive oral rehydration therapy according to the investigator's standard of care

Attend up to 4 clinic visits over 5 days and receive 4 follow-up phone calls

Provide blood samples on Day 1 and Day 3 for pharmacokinetic testing (rifaximin group only)

Provide stool samples to identify bacterial pathogens

Keep a diary of stool frequency and consistency to help determine when diarrhea resolves

Be monitored for side effects, vital signs, and laboratory changes

DETAILED DESCRIPTION:
This study is a randomized, open-label clinical trial designed to evaluate the pharmacokinetics, safety, and efficacy of rifaximin 200 mg in pediatric participants aged 6 to 11 years with acute diarrhea of suspected bacterial etiology. Acute diarrhea may be caused by bacterial infections such as E. coli, Shigella, Salmonella, or Campylobacter.

Participants are randomly assigned to receive either rifaximin 200 mg plus oral rehydration therapy (ORT) or ORT alone. Participants in the rifaximin group take one tablet three times a day for 3 days, in addition to ORT according to the investigator's standard of care. Participants in the ORT-alone group receive ORT only.

The primary objective is to assess how rifaximin is absorbed, distributed, and eliminated in children (pharmacokinetics). Secondary objectives include evaluating the safety and tolerability of rifaximin and assessing whether rifaximin plus ORT helps resolve diarrhea faster than ORT alone.

Safety assessments include monitoring adverse events, vital signs, and laboratory tests (hematology, chemistry, and urinalysis). Participants or their caregivers keep a daily diary to record stool frequency and consistency, time to last unformed stool, and any related symptoms such as abdominal cramps, nausea, vomiting, or flatulence. Stool samples are collected to identify the bacterial pathogen(s) causing diarrhea.

Pharmacokinetic assessments are conducted in participants receiving rifaximin plus ORT, with blood samples collected on Day 1 and Day 3: pre-dose, 1 hour post-dose, and 8 hours post-dose. Plasma samples are analyzed for rifaximin and 25-desacetyl rifaximin to determine pharmacokinetic parameters, including maximum concentration (Cmax), time to maximum concentration (Tmax), and area under the concentration-time curve (AUC).

Participants attend up to four clinic visits over the 5-day study period and receive follow-up phone calls on Days 6, 7, 8, and 30 to monitor safety and collect diary information. Compliance with study drug and ORT administration is assessed throughout the study.

This study is designed to provide information on rifaximin pharmacokinetics, its safety in children, and the potential benefit of rifaximin plus ORT in resolving acute diarrhea of suspected bacterial origin.

ELIGIBILITY:
Inclusion Criteria:

1. Consent and assent are appropriately obtained prior to any study related activities, including discontinuation of any prohibited medications (subjects must sign an assent for the study and a parent or a legal guardian must sign the informed consent).
2. Subject is between 6 to 11 (and 11 months) years of age, inclusive, and weighs at least 15 kg (33 lbs) at Screening.
3. Females of childbearing (reproductive) potential must have a negative urine and serum pregnancy test at Screening and agree to use a highly effective method of contraception throughout their participation in the study. Acceptable methods of contraception are those alone or in combination, that result in a low failure rate (ie, less than 1% per year) when used consistently and correctly and include hormonal methods (oral, injected or implanted), intrauterine device or intrauterine system or double barrier methods (simultaneous use of a physical barrier method by the subject and male partner, including a male condom and an occlusive cap [diaphragm or cervical/vault cap] with spermicidal). Abstinence or partner(s) with a vasectomy may be considered an acceptable method of contraception at the discretion of the Investigator.

   NOTE: Female subjects are considered of child-bearing potential if they are (a) physiologically capable of becoming pregnant, defined as a female who has experienced menarche and (b) they will be, or could possibly be, engaging in sexual activity during the course of the study.
4. Subject has diarrhea of suspected bacterial etiology defined by:

   * At least 3 unformed stools in the last 24 hours prior to Screening.
   * A fever ≥ 100.4°F (38°C) and ≤ 102.2°F (39°C) or has had a fever of ≥ 100.4°F (38°C) and ≤ 102.2°F (39°C) at any time since the development of abdominal pain or diarrhea.
   * Illness for less than 96 hours at Screening.
5. Parent or legal guardian and subject, when applicable based on aged, are capable of understanding the requirements of the study and willing to comply with all study procedures and visits.

Exclusion Criteria:

1. Subject has a history of chronic diarrhea.
2. Subject is unable to eat or drink.
3. Subject has at least one of the following signs or symptoms:

   * Presence of fever >39°C (>102.2°F).
   * Presence of frank blood in stool.
4. Subject has taken >2 doses of anti-diarrheal therapies in the 24 hours prior to randomization.
5. Subject has taken any oral antimicrobial drug within 14 days of randomization.
6. Subject has an unstable medical condition, in the opinion of the Investigator, (including, but not limited to, evidence of severe dehydration noted by tachycardia, abnormal blood pressure, or decreased skin turgor) at the Screening visit.
7. Subject has known, clinically significant hepatic disease manifested by twice the age and sex-adjusted upper limit of normal (2 × ULN) for any of the following liver function tests: alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transferase, alkaline phosphatase, or total bilirubin (except in isolated elevation of unconjugated bilirubin).
8. Subject has known, clinically significant renal disease (eg, 1.5 × ULN of serum creatinine or 2 × ULN of blood urea nitrogen levels).
9. Subject has serum sodium of ≥150 mEq/L and serum potassium ≤3.0 mEq/L.
10. Subject has a known hypersensitivity or allergy to Xifaxan®, rifampin, rifamycin-derived antibiotics, or any of the components of the rifaximin (Xifaxan®) formulations used in this study.
11. Subject is pregnant or lactating or plans to become pregnant during the study.
12. Subject has had a previous history of malignancy.
13. Subject has a history of tuberculosis infection and/or has received treatment for tuberculosis infection.
14. Subject has any concurrent illness, disability or circumstance that may affect the interpretation of clinical data, could cause noncompliance with treatment or visits or otherwise contraindicates participation in this study in the opinion of the Investigator.
15. Subject has had significant blood loss within the 30 days prior to the Screening visit which prevents the collection of the blood volume required for this study.
16. Subject has participated in an investigational drug or device study within the 30 days prior to randomization.
17. Subject's parent or legal guardian, or an immediate family member is an employee of the site that is directly involved in the management, administration, or support of this study.
18. Subject and/or legal guardian is unwilling or unable to comply with the study protocol for any other reason.
19. Subject has a serum glucose level at screening that deviates from the reference range established by the central laboratory.
20. Subject is taking a concomitant medication that is a P-glycoprotein (P-gp) inhibitor.
21. Subject is taking warfarin for a pre-existing condition.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2027-04-20 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of Rifaximin | Days 1 and 3
  Cmax levels following rifaximin 200 mg + ORT
Time to Maximum Plasma Concentration (Tmax) of Rifaximin | Days 1 and 3
  Tmax for rifaximin following rifaximin 200 mg + ORT
Area Under the Plasma Concentration-Time Curve From Time 0 to Last Quantifiable Concentration (AUC0-last) for Rifaximin | Days 1 and 3
  Area under the concentration-time curve to last measurable concentration
Area Under the Plasma Concentration-Time Curve Over the Dosing Interval (AUC0-τ) for Rifaximin | Days 1 and 3
  Area under the concentration-time curve over the dosing interval
Proportion of participants with Clinical Cure | Up to Day 5 (End of Treatment)
  Proportion of participants achieving clinical cure, defined as either:
  1. No unformed stools within a 48-hour period with no fever (with or without other clinical symptoms such as abdominal cramps or pain, excess gas/flatulence, nausea, vomiting, urgency, tenesmus); or
  2. No watery stools and no more than two soft stools within a 24-hour period with no fever and no other clinical symptoms except for mild excess gas/flatulence.

SECONDARY OUTCOMES:
Time to Last Unformed Stool (TLUS) | Up to Day 5 (End of Treatment)
  Time in hours from the first dose of study treatment to the last unformed stool, after which clinical cure is declared, based on subject/caregiver diary entries.
Incidence of Treatment-Emergent Adverse Events (AEs) | Day 1-30
  Number and percentage of participants with AEs and SAEs
Change From Baseline in Clinical Laboratory Parameters | Day 1-30
  Changes in hematology, chemistry, and urinalysis values
Change From Baseline in Vital Signs | Day 1-30
  Change in temperature, blood pressure, and pulse

OTHER OUTCOMES:
Detection of Bacterial Pathogens in stool samples | Screening (Day -2 to Day 1)
  Identification of bacterial pathogen(s) isolated from stool samples of enrolled participants.

IPD SHARING:
Plan to Share IPD: No
The sponsor does not intend to share individual participant-level data from this study. Summary results will be posted in accordance with applicable regulations.